CLINICAL TRIAL: NCT00764868
Title: A Phase III, Open-Label, Extension, Multi-Center, Safety and Efficacy Study of Lisdexamfetamine Dimesylate (LDX) in Adolescents Aged 13-17 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Vyvanse Adolescent Open-Label Safety and Efficacy Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPD489-306
Record Dates: First submitted 2008-09-29; First posted 2008-10-02 (Estimated); Results first posted 2011-03-28 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDX (Experimental): Lisdexamfetamine Dimesylate (LDX)
  Interventions: Drug: Lisdexamfetamine Dimesylate (LDX)

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate (LDX) — optimal dose of 30, 50 or 70 mg once daily
  Other Names: Vyvanse

SUMMARY:
The primary objective of this study is to evaluate the long-term safety of LDX administered as a daily morning dose (30, 50, and 70 mg/day) in the treatment of adolescents (13-17 years of age inclusive at the time of consent).

DETAILED DESCRIPTION:
Not Required

ELIGIBILITY:
Inclusion

1. Subject is a male or female aged 13-17 years inclusive at the time of consent of the antecedent study (SPD489-305).
2. Subject satisfied all entry criteria for the antecedent study (SPD489-305), and completed a minimum of 3 weeks of double-blind treatment and reached Visit 3 of the antecedent study (SPD489-305), without experiencing any clinically significant adverse events (AEs) that would preclude exposure to LDX.

Exclusion

1. Subject was terminated from SPD489-305 for non-compliance and/or experienced a serious adverse event (SAE) or AE resulting in termination from the antecedent study (SPD489-305).
2. Subject has a current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as any severe comorbid Axis II disorder or severe Axis I disorder (such as Post Traumatic Stress Disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder) or other symptomatic manifestations, such as agitated states, marked anxiety, or tension that, in the opinion of the examining clinician, will contraindicate treatment with LDX or confound efficacy or safety assessments. Comorbid psychiatric diagnoses will be established at the Screening Visit (Visit -1) of the antecedent study (SPD489-305) with the Screening interview of the Kiddie-SADS-Present and Lifetime - Diagnostic Interview (K-SADS-PL) and additional modules if warranted by the results of the initial interview. Participation in behavioral therapy, provided the subject was receiving the therapy for at least 1 month at the time of the Baseline Visit (Visit 0) of the antecedent study (SPD489-305).
3. Subject has a conduct disorder. Oppositional Defiant Disorder is not exclusionary.
4. Subject is currently considered a suicide risk, has previously made a suicide attempt or has a prior history of, or is currently demonstrating suicidal ideation.
5. Subject is underweight based on Center for Disease Control and Prevention Body Mass Index (BMI)-for-age gender specific charts at the Enrollment Visit (Visit 1) of this study. Underweight is defined as a BMI < 5th percentile.
6. Subject has a concurrent chronic or acute illness or unstable medical condition that could confound the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol.
7. Subject has a history of seizures (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder.
8. Subject has a known history symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
9. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
10. Subject has any clinically significant ECG, based on the Principal Investigator's judgment, at Visit 4/ET of the antecedent study (SPD489-305).
11. Subject is taking any medication that is excluded.
12. Subject has a documented allergy, hypersensitivity or intolerance to amphetamine.
13. Subject has a recent history (within the past 6 months) of suspected substance abuse or dependence disorder (excluding nicotine) in accordance with DSM-IV-TR criteria.
14. Subject has glaucoma.
15. Subject is taking other medications that have central nervous system (CNS) effects or affect performance, such as sedating antihistamines and decongestant sympathomimetics, or are monoamine oxidase inhibitors. Stable use of bronchodilator inhalers is not exclusionary.
16. Subject is female and is pregnant or lactating.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 269 (Actual)
Dates: Start 2008-11-13 (Actual); Primary Completion 2010-04-22 (Actual); Study Completion 2010-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (45):
- United States (45):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Valley Clinical Research, Inc., El Centro, California
  - Penninsula Research Associates, Inc., Rolling Hills Estates, California
  - Psychiatric Centers at San Diego (PCSD-Feighner Research Institute), San Diego, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Amedica Research Institute, Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Clinco Inc., Terre Haute, Indiana
  - CIENTIFICA, Inc. at Prairie View, Newton, Kansas
  - Psychiatric Associates, Overland Park, Kansas
  - Vince and Associates Clinical Research, Inc., Overland Park, Kansas
  - Pedia Research LLC., Owensboro, Kentucky
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Bart Sangal, Troy, Michigan
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Children's Specialized Hospital, Toms River, New Jersey
  - Bioscience Research, LLC, Mount Kisco, New York
  - Triangle Neuropsychiatry, PLLC, Durham, North Carolina
  - Innovis Health/Odyssey Research, Fargo, North Dakota
  - University Hospitals of Cleveland Division of Child & Adolescent Psychiatry, Cleveland, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - OCCI, Eugene, Oregon
  - Summit Research Network, Portland, Oregon
  - OCCI, INC (Oregon Center for Clinical Investigations, Inc.), Salem, Oregon
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Youth and Family Research Program/WPIC ADHD Research Program, Pittsburgh, Pennsylvania
  - CNS Healthcare, Memphis, Tennessee
  - Future Search Trials, Austin, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Red Oak Psychiatry Associates P.A., Houston, Texas
  - ADHD Clinic of San Antonio, San Antonio, Texas
  - Vermont Clinical Study Center, Burlington, Vermont
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Neuroscience, Inc., Herndon, Virginia
  - Dominion Clinical Research, Midlothian, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Result] Findling RL, Cutler AJ, Saylor K, Gasior M, Hamdani M, Ferreira-Cornwell MC, Childress AC. A long-term open-label safety and effectiveness trial of lisdexamfetamine dimesylate in adolescents with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2013 Feb;23(1):11-21. doi: 10.1089/cap.2011.0088. PMID 23410138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects had to have satisfied all entry criteria for the antecedent study (SPD489-305, NCT00735371) and completed a minimum of 3 weeks of double-blind treatment and reached Visit 3 of the antecedent study (SPD489-305), without experiencing any clinically significant adverse events that would preclude exposure to LDX.
Pre-assignment Details: 269 subjects were enrolled, but 4 were not dosed during the study and thus excluded from the Safety Population.
Groups:
- Lisdexamfetamine Dimesylate (LDX): Subjects who received either Lisdexamfetamine Dimesylate (LDX) or placebo during antecedent study 489-305 were eligible for 489-306. All subjects were titrated to their optimal dose of LDX (30, 50 or 70 mg per day).
Period: Overall Study
Arm/Group | Lisdexamfetamine Dimesylate (LDX)
Started | 269
Completed | 156
Not Completed | 113
Not completed — Adverse Event | 18
Not completed — Withdrawal by Subject | 31
Not completed — Non-compliance | 16
Not completed — Lost to Follow-up | 25
Not completed — Lack of Efficacy | 5
Not completed — Subject moved | 7
Not completed — Pregnancy | 3
Not completed — Prohibited medication | 1
Not completed — Out of town | 1
Not completed — Misuse and compliance of study drug | 1
Not completed — Subject sent to boarding school | 1
Not completed — Met an exclusion criteria | 1
Not completed — Positive drug screen | 2
Not completed — Sponsor requested withdrawal | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lisdexamfetamine Dimesylate (LDX)
Number analyzed (Participants) | 265
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics were calculated from the Safety Population (n = 265) defined as all randomized subjects who received at least 1 dose of investigational product. Baseline and demographic characteristics are calculated from entry into the antecedent study (SPD489-305, NCT00735371).
  years | 14.5 (1.30)
Age, Customized [Count of Participants; unit: Participants]
  13 to 14 years | 144
  15 to 17 years | 121
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 187
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 265

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (From the Antecedent Study, SPD489-305) in the Attention-Deficit/Hyperactivity Disorder Rating Scale, Fourth Edition (ADHD-RS-IV) Total Score at up to 52 Weeks
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and up to 52 weeks
Population: Full Analysis Set (FAS) defined as all subjects who took at least 1 dose of investigational product and have a valid baseline and at least 1 valid follow-up assessment of the primary outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX)
Number analyzed (Participants) | 265
Units on a scale | -26.2 (9.75)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX); Test type: Superiority or Other; p < 0.001, t-test, 2 sided; t-test of LDX at baseline and 52 weeks

2. Secondary Outcome: Percent of Participants With Improvement in Clinical Global Impression-Improvement (CGI-I)
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: up to 52 weeks
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX)
Number analyzed (Participants) | 265
Percent of participants | 87.2

3. Secondary Outcome: Change From Baseline (From the Antecedent Study, SPD489-305) in the Youth Quality of Life Instrument-Research Version (YQOL-R) Total Score at up to 52 Weeks
Description: The Youth Quality of Life-research version (YQOL-R) is a validated 56-item generic instrument for comparing quality of life of adolescents across condition groups that scores each question on a scale from 0 (never) to 4 (very often). The YQOL scores are transformed to a 0-100 scale for easy interpretability. Higher scores indicate better quality of life.
Time Frame: Baseline and Up to 52 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX)
Number analyzed (Participants) | 237
Units on a scale | 3.9 (9.73)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX); Test type: Superiority or Other; p < 0.001, t-test, 2 sided; t-test of LDX at baseline and 52 weeks

ADVERSE EVENTS:
Description: Safety population is defined as all subjects who take at least 1 dose of investigational product. In the Serious Adverse Events, the same subject reported multiple adverse events.
Arm/Group | Lisdexamfetamine Dimesylate (LDX)
Serious Adverse Events (participants affected / at risk) | 10/265
Other Adverse Events (participants affected / at risk) | 230/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine Dimesylate (LDX) (N=265)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 3 (4)
Syncope Vasovagal (Nervous system disorders) | 1 (1)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Aggression (Psychiatric disorders) | 2 (2)
Testicular Torsion (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine Dimesylate (LDX) (N=265)
Dry Mouth (Gastrointestinal disorders) | 14 (15)
Irritability (General disorders) | 33 (36)
Influenza (Infections and infestations) | 18 (18)
Nasopharyngitis (Infections and infestations) | 19 (26)
Upper Respiratory Tract Infection (Infections and infestations) | 58 (74)
Weight Decreased (Investigations) | 43 (46)
Decreased Appetite (Metabolism and nutrition disorders) | 56 (71)
Dizziness (Nervous system disorders) | 14 (16)
Headache (Nervous system disorders) | 55 (81)
Insomnia (Psychiatric disorders) | 32 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.